CLINICAL TRIAL: NCT07244627
Title: Anaesthetic Technique for Minor Lower Limb Amputation Surgery (ATLLAS): A Retrospective Review of Outcomes
Brief Title: Anaesthetic Technique for Minor Lower Limb Amputation Surgery (ATLLAS)
Acronym: ATLLAS
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 338872
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia; Amputation; Traumatic, Leg, Lower

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Major lower limb amputation is recognised as a significant cause of morbidity and mortality. In the United Kingdom, 30-day in-hospital mortality is up to 8.7%. Minor lower limb amputations, defined as amputation at or below the ankle, are often considered minor procedures, but mortality at one month is 3.5%, similar to that of below knee amputations and 20% at one year. Any amputation is an indicator of poor health and should be considered a pivotal event in a patient's healthcare journey. In England alone, 21,738 minor lower limb amputations were performed between 2017 and 2020, with annual procedures on an increasing trajectory. Recent work has demonstrated striking regional differences in rates of major lower limb amputations in England which the authors ascribed to inequalities in the provision of healthcare. Improving the regional provision of support services for amputees is also part of the current governments NHS Long Term Workforce Plan (https://lordslibrary.parliament.uk/access-to-prosthetics-for-amputees-in-england/).

While multiple studies have aimed to assess the impact of anaesthetic technique on outcomes following major lower limb amputation, there is little published data on factors impacting morbidity and mortality following minor lower limb amputation surgery. Evidence from the USA has shown deleterious effect of general anaesthesia (GA) as compared to regional anaesthesia for minor lower limb amputation in patients with peripheral artery disease. Higher rates of post-operative wound disruption, pneumonia, prolonged intubation, and septic shock were demonstrated with general anaesthesia rather than regional anaesthesia.

Investigators have performed a single centre retrospective review of 382 patients undergoing minor lower limb amputation for vascular disease in our Trust (UHNM). We found that our patients undergoing these procedures under peripheral nerve block (PNB) techniques were older with higher rates of heart and kidney disease than those receiving a general anaesthetic. Despite this, these patients had reduced complications and length of hospital stay than the fitter patients. The difference seen here became even more pronounced following propensity matching. Investigators demonstrated a clinically significant reduction in the respiratory complication rate of 5.3% and overall complication rate of 12% and a reduction in length of stay of 6 days following use of peripheral nerve blocks rather than general anaesthesia. Investigators also demonstrated a reduction in length of stay of 4 days when DARF Form v4 - July 2023 16 administering peripheral nerve blocks rather than neuraxial anaesthesia (NA). This small and monocentric study suggests that there is value in repeating this process in a larger, national dataset.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 and over).
* National Vascular Registry data field - Procedure undertaken - amputation through ankle or below.
* Procedure undertaken between 1st January 2019 and 1st January 2025.

Exclusion Criteria:

* Amputations due to trauma, neurological disease or chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the National Vascular Registry (NVR) database for minor lower limb amputations undertaken between January 2019 and January 2025.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Morbidity following amputation | 30 days post amputation
  Compare all cause morbidity at 30 days following amputation under general, neuraxial and peripheral nerve block anaesthesia, converting it from local to national data

SECONDARY OUTCOMES:
Comparing emergency and elective outcomes | 30 days post amputation
  Comparing emergency and elective outcomes against American society of Anaesthesiologists (ASA) grading. ASA classification uses a grading system of I (one) through V (five), with I identifying a person in good health and V as a person with a severe, life-threatening condition. The sixth (VI) status identifies deceased organ donors.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of North Midlands, Stoke-on-Trent, Staffordshire, United Kingdom

REFERENCES:
- [Background] Yammine K, Hayek F, Assi C. A meta-analysis of mortality after minor amputation among patients with diabetes and/or peripheral vascular disease. J Vasc Surg. 2020 Dec;72(6):2197-2207. doi: 10.1016/j.jvs.2020.07.086. Epub 2020 Aug 21. PMID 32835790
- [Background] Ahmad N, Thomas GN, Gill P, Chan C, Torella F. Lower limb amputation in England: prevalence, regional variation and relationship with revascularisation, deprivation and risk factors. A retrospective review of hospital data. J R Soc Med. 2014 Dec;107(12):483-9. doi: 10.1177/0141076814557301. Epub 2014 Nov 11. PMID 25389229
- [Background] Chery J, Semaan E, Darji S, Briggs WT, Yarmush J, D'Ayala M. Impact of regional versus general anesthesia on the clinical outcomes of patients undergoing major lower extremity amputation. Ann Vasc Surg. 2014 Jul;28(5):1149-56. doi: 10.1016/j.avsg.2013.07.033. Epub 2013 Dec 14. PMID 24342828
- [Background] Waton S, Johal A, Birmpili P et al. National Vascular Registry: 2022 Annual Report. London: The Royal College of Surgeons of England, November 2022
- [Background] Khan SA, Qianyi RL, Liu C, Ng EL, Fook-Chong S, Tan MG. Effect of anaesthetic technique on mortality following major lower extremity amputation: a propensity score-matched observational study. Anaesthesia. 2013 Jun;68(6):612-20. doi: 10.1111/anae.12182. Epub 2013 Apr 1. PMID 23550809
- [Background] Pisansky AJB, Brovman EY, Kuo C, Kaye AD, Urman RD. Perioperative Outcomes after Regional Versus General Anesthesia for Above the Knee Amputations. Ann Vasc Surg. 2018 Apr;48:53-66. doi: 10.1016/j.avsg.2017.10.014. Epub 2017 Dec 5. PMID 29217448
- [Background] Walsh M, Lim S, Gill L, et al. Deleterious Effects of General Anesthesia on Minor Foot Amputations. Abstract from the 2018 Midwestern Vascular Surgical Society Annual Meeting, Journal of Vascular Surgery 2018; 68: E54-55
- See also: Related Info — https://fingertips.phe.org.uk/static-reports/diabetes-footcare/national-diabetic-footcare-report.html